CLINICAL TRIAL: NCT04668248
Title: Novel Application of Simulation for Providers to Overcome Decisional Gaps in High-risk Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Ideas42 (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julie Lauffenburger, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020P003643; 5P30AG064199-02 (NIH)
Record Dates: First submitted 2020-11-19; First posted 2020-12-16 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Medication Administered in Error; Antipsychotics and Neuroleptics Toxicity
Keywords: Simulation; Behavioral principles; Drug; Education; Pharmacology; Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation intervention (Experimental): Providers assigned to the intervention arm will participate in a short simulation training at the beginning of their 2-week block (planned for their second day). The training will take place at the Neil and Elise Wallace STRATUS Center for Medical Simulation at Brigham and Women's Hospital and will follow all of their recommended and hospital-recommended practices on social distancing, including the learning limits.
  Interventions: Other: Simulation
- Online education intervention (Active Comparator): Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines.
  Interventions: Other: Online educational training

INTERVENTIONS:
Other: Simulation — The simulation will consist of a one-time, short immersive simulation session at the STRATUS Center for Medical Education at BWH. The session will be conducted for up to one intern at the same time, in accordance with social distancing practices at BWH. This simulation session will consist of one short, hands-on scenario of simulated patient experiences with expert facilitators in the simulated hospital rooms to help providers identify when they are in the hot state and their reactions, and work on improving communication skills, differential diagnoses, and alternative therapeutic options. These scenarios are intended to simulate both in-person and virtual interactions that are common in the inpatient setting. During these trainings, we will use behavioral principles like time pressure and increasing cognitive load to simulate a "hot state" environment. After the scenarios, the facilitator will perform a debriefing session for the interns.
  Arms: Simulation intervention
Other: Online educational training — Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines. This information will be in the form of electronically-delivered links to information already housed and available at BWH, including reviewing BWH guidelines and literature about transfusion reactions. The interns will be asked to answer several clinical questions about optimal prescribing. Albumin and related products are also high-risk medications often overprescribed on twilight shifts.
  Arms: Online education intervention

SUMMARY:
This pilot project aims to reduce the prescribing of high-risk medications, such as antipsychotics and benzodiazepines, to hospitalized older adults. To accomplish this, this project consists of two phases. The purpose is to determine whether a novel simulation-based training program reduces prescribing of suboptimal medications for older adults. A 2-arm pilot randomized controlled trial will be conducted to test a simulation-based, principle-driven intervention targeting high-risk prescribing practices versus control.

DETAILED DESCRIPTION:
The overarching goal is to determine whether a newly-designed simulation-based training program for providers based on underlying principles of System 1 and System 2 thinking reduces prescribing of high-risk medications for hospitalized older adults versus control, with the ultimate goal of improving patient safety. Subsequent prescribing for patients cared for by other providers and other adoption and implementation outcomes will be measured to explore the extent to which the intervention could be used at scale.

36 interns practicing on the general medicine inpatient service at Brigham and Women's Hospital will be assigned to the "twilight" team. Interns who consent will be randomized in a 1:1 ratio to one of 2 arms: (a) Arm 1: simulation training and (b) Arm 2: control (online educational training).

Patients who will be included in the analysis will include adults ≥65 years old who are admitted to the BWH/BWFH general medicine service under the care of one of the consenting interns (specifically, with the intern listed as the "Responding Clinician")

ELIGIBILITY:
Residents and interns at Brigham and Women's Hospital will be eligible for this trial if they care for older adults (age 65+) admitted to one of the general medicine wards during an evening shift.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lauffenburger JC, DiFrancesco MF, Bhatkhande G, Crum KL, Kim E, Robertson T, Oran R, Hanken KE, Haff N, Coll MD, Avorn J, Choudhry NK. Pragmatic trial evaluating the impact of simulation training on high-risk prescribing to older adults by junior physicians. J Am Geriatr Soc. 2024 May;72(5):1420-1430. doi: 10.1111/jgs.18862. Epub 2024 Mar 8. PMID 38456561
- [Derived] Lauffenburger JC, DiFrancesco MF, Barlev RA, Robertson T, Kim E, Coll MD, Haff N, Fontanet CP, Hanken K, Oran R, Avorn J, Choudhry NK. Overcoming Decisional Gaps in High-Risk Prescribing by Junior Physicians Using Simulation-Based Training: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 27;11(4):e31464. doi: 10.2196/31464. PMID 35475982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First-year medical resident physicians (i.e., interns) who provide care on inpatient general medicine services at Brigham and Women's Hospital from March to December 2021 were eligible for this trial if they were assigned to one of the general medicine wards and were scheduled for twilight rotations.
Groups:
- Simulation Intervention: Providers assigned to the intervention arm will participate in a short simulation training at the beginning of their 2-week block (planned for their second day). The training will take place at the Neil and Elise Wallace STRATUS Center for Medical Simulation at Brigham and Women's Hospital and will follow all of their recommended and hospital-recommended practices on social distancing, including the learning limits.
  Simulation: The simulation will consist of a one-time, short immersive simulation session at the STRATUS Center for Medical Education at BWH. This simulation session consisted of a short hands-on scenario of simulated patient experiences with expert facilitators in the simulated hospital rooms to help providers identify when they are in the hot state and their reactions, and work on improving communication skills, differential diagnoses, and alternative therapeutic options. This scenario was intended to simulate both in-person and virtual interactions that are common in the inpatient setting. During these trainings, we used behavioral principles like time pressure and increasing cognitive load to simulate a "hot state" environment. After the scenarios, the facilitator performed a debriefing session for the interns.
- Online Education Intervention (Control): Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines.
  Online educational training: Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines. This information will be in the form of electronically-delivered links to information already housed and available at BWH, including reviewing BWH guidelines and literature about transfusion reactions. The interns will be asked to answer several clinical questions about optimal prescribing. Albumin and related products are also high-risk medications often overprescribed on twilight shifts. Receiving education about another high-risk medication will reduce contamination and allow the ability to measure outcomes to other high-risk medications.
Period: Overall Study
Arm/Group | Simulation Intervention | Online Education Intervention (Control)
Started | 24 | 23
Sick | 1 | 0
Schedule Change | 4 | 0
Did Not Complete Training in Time | 0 | 2
Completed | 19 | 21
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simulation Intervention | Online Education Intervention (Control) | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (2.3) | 29.0 (2.5) | 28.4 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 8 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 15 | 24
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 1 | 4
Clinical Service Type, N(%) [Count of Participants; unit: Participants]
  General Medicine Service | 9 | 9 | 18
  Integrated Teaching Unit | 7 | 10 | 17
  Faulkner General Medicine Service | 3 | 2 | 5
Department, N (%) [Count of Participants; unit: Participants]
  Medicine | 12 | 13 | 25
  Other | 7 | 8 | 15
Stage of Training, N(%) [Count of Participants; unit: Participants]
  May-June 2021 | 5 | 7 | 12
  Sept-Dec 2021 | 14 | 14 | 28
Survey Responses, mean (SD) [Mean (Standard Deviation); unit: units on a scale]
  Baseline State-Trait Anxiety Inventory (STAI)-6 Score, range 0-63 (higher is more anxiety) | 14.9 (3.2) | 15.1 (3.8) | 15.0 (3.5)
  Baseline Reactions to Uncertainty Score, range 8-32 (higher is more certain) | 26.9 (8.5) | 28.8 (8.5) | 27.9 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: High-risk Medication Doses
Description: This will include the number of pills or injection order of high-risk medications (i.e., anti-psychotics, benzodiazepines, and sedative hypnotic "Z-drugs") administered to eligible patients (i.e., those 65 or older not previously on one of these medications)
Time Frame: Within 2-week service block of participating provider
Population: The analysis was conducted among patients of these providers who meet eligibility criteria for inclusion in the analysis (n=522 total).
Measure: Mean (Standard Deviation); unit: No. of med orders by patient per intern
Groups:
- Simulation Intervention: Providers assigned to the intervention arm will participate in a short simulation training at the beginning of their 2-week block (planned for their second day). The training will take place at the Neil and Elise Wallace STRATUS Center for Medical Simulation at Brigham and Women's Hospital and will follow all of their recommended and hospital-recommended practices on social distancing, including the learning limits.
  Simulation: The simulation will consist of a one-time, short immersive simulation session at the STRATUS Center for Medical Education at BWH. The session will be conducted for up to 4 interns at the same time, in accordance with social distancing practices at BWH. This simulation session will consist of 2 short, hands-on scenarios of simulated patient experiences with expert facilitators in the simulated hospital rooms to help providers identify when they are in the hot state and their reactions, and work on improving communication skills, differential diagnoses, and alternative therapeutic options. These scenarios are intended to simulate both in-person and virtual interactions that are common in the inpatient setting. During these trainings, we will use behavioral principles like time pressure and increasing cognitive load to simulate a "hot state" environment. After the scenarios, the facilitator will perform a debriefing session for the interns.
- Online Education Intervention: Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines.
  Online educational training: Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines. This information will be in the form of electronically-delivered links to information already housed and available at BWH, including reviewing BWH guidelines and literature about transfusion reactions. The interns will be asked to answer several clinical questions about optimal prescribing. Albumin and related products are also high-risk medications often overprescribed on twilight shifts. Receiving education about another high-risk medication will reduce contamination and allow the ability to measure outcomes to other high-risk medications.
Arm/Group | Simulation Intervention | Online Education Intervention
Number analyzed (Participants) | 259 | 263
No. of med orders by patient per intern
  All orders | 0.049 (0.25) | 0.052 (0.27)
  Standing orders | 0.036 (0.22) | 0.019 (0.16)
  PRN orders | 0.013 (0.11) | 0.032 (0.18)
  One-time orders | 0.030 (0.02) | 0.013 (0.11)

2. Secondary Outcome: Percentage of Patients Discharged With Inappropriate Medications
Description: Percentage of patients discharged with inappropriate medications, measured through electronic health record data
Time Frame: 2 week follow-up period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Online Education Intervention (Control): Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines.
  Online educational training: Providers assigned to the control arm received online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines. This information were in the form of electronically-delivered links to information already housed and available at BWH, including reviewing BWH guidelines and literature about transfusion reactions. The interns were asked to answer several clinical questions about optimal prescribing. Receiving education about another high-risk medication was designed to reduce contamination and allow the ability to measure outcomes to other high-risk medications.
Arm/Group | Simulation Intervention | Online Education Intervention (Control)
Number analyzed (Participants) | 259 | 263
Participants | 27.0 | 20.0

3. Other Pre Specified Outcome: Number and Percentage of Participants Signing Consent Forms
Description: Percentage of consenting providers out of those eligible (measured by the Amion scheduling system)
Time Frame: Between study initiation and end of recruitment up to 10 months
Population: The denominator for this analysis is the number of providers who were contacted for participation in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Study Population: Providers were first screened for eligibility and then invited to participated. Once consent was provided, they were randomized to intervention or control. The denominator for this outcome therefore is the number of providers who were screened as potentially eligible.
Arm/Group | Eligible Study Population
Number analyzed (Participants) | 97
Participants | 48

4. Other Pre Specified Outcome: Rate of Simulation or Online Educational Training Completion
Description: Rate of simulation training completion or online educational training completion
Time Frame: 2 week follow-up period
Population: Number of providers who were randomized to the study and completed the training (n=47 were randomized appropriately).
Measure: Count of Participants; unit: Participants
Groups:
- Online Education Intervention: Providers assigned to the control arm will receive online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines.
  Online educational training: Providers assigned to the control arm received online educational training about other poorly-prescribed medications, including albumin, transfusion, and blood product repletion guidelines. This information were in the form of electronically-delivered links to information already housed and available at BWH, including reviewing BWH guidelines and literature about transfusion reactions. The interns were asked to answer several clinical questions about optimal prescribing. Receiving education about another high-risk medication was designed to reduce contamination and allow the ability to measure outcomes to other high-risk medications.
Arm/Group | Simulation Intervention | Online Education Intervention
Number analyzed (Participants) | 24 | 23
Participants | 19 | 21

5. Other Pre Specified Outcome: Feedback and Issues Reported by the Interns or Study Staff
Description: Feedback and issues reported by the interns or study staff (measured in the endline questionnaire)
Time Frame: Between study initiation and end of recruitment up to 10 months
Population: Interns randomized to the study and provided data in the endline questionnaire. No feedback or issues were reported in the endline questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Simulation Intervention | Online Education Intervention (Control)
Number analyzed (Participants) | 19 | 21
Participants | 0 | 0

6. Other Pre Specified Outcome: Satisfaction With the Intervention
Description: Satisfaction with the intervention (measured in the endline questionnaire). This item was measured using several validated questions. The final summary question is used to summarize satisfaction, with the percentage of those strongly agreeing with the statement that "I learned new information during participation in the study that I would not have learned otherwise" shown by each arm below.
Time Frame: 2 week follow-up period
Population: Providers who completed the endline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Simulation Intervention | Online Education Intervention (Control)
Number analyzed (Participants) | 19 | 21
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: Adverse events for provider participants were collected from the beginning of randomization until the end of their 2-week follow-up.
Arm/Group | Simulation Intervention | Online Education Intervention (Control)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT04668248/Prot_SAP_000.pdf